CLINICAL TRIAL: NCT02401568
Title: Morphologic and Biomechanical Analysis of the Carpal Ligaments: a Kinematic Study on Dynamic Area Detector CT
Brief Title: Morphologic and Biomechanical Analysis of the Carpal Ligaments
Acronym: EDLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A00845-42
Record Dates: First submitted 2015-03-11; First posted 2015-03-30 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2020-07

CONDITIONS: Joint Instability; Wrist Injuries
MeSH Terms: conditions — Joint Instability; Wrist Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal subjects (Other): No morphologic changes in carpal ligaments or clinical signs of wrist instability.
  Dynamic CT of the wrist will be performed before and after arthrography.
  Interventions: Device: Dynamic CT; Procedure: Arthrography
- Wrist instability (Other): Morphologic ligament changes (e.g. partial or complete rupture) Dynamic CT of the wrist will be performed before and after arthrography.
  Interventions: Device: Dynamic CT; Procedure: Arthrography

INTERVENTIONS:
Device: Dynamic CT — Various low dose CT acquisitions will be successively performed on the wrist to allow a four dimensional evaluation. The same type of acquisition will be performed during various manoeuvers (radio-ulnar deviation, clenching fist, and dart-throwing motion).
Procedure: Arthrography — percutaneous intra-articular injection of contrast media in the medio-carpal and radio-carpal joints

SUMMARY:
Compare various dynamic biomechanical markers (distances and angles) in the wrist during dynamic CT studies in three groups of patients: Normal subjects, with scapholunate instability and with other types of wrist instability.

DETAILED DESCRIPTION:
Patients referred for the evaluation of wrist pain with CT arthrography will be eligible for inclusion. Patients will benefit from dynamic CT acquisitions before and after arthrography with three maneuvers: radio-ulnar deviation, clenching fist and dart throwing motion. Patients will also benefit from a wrist MR study on a 3 tesla scanner.

The morphology of the carpal ligaments will be evaluated on static imaging (MR and CT arthrograph) and on dynamic CT arthrography.

Distance and angular measurements will be obtained from dynamic CT studies using an appropriate post processing tool (4D-Ortho).

Data obtained with dynamic wrist evaluation will be correlated to ligament morphology, classical wrist instability criteria on conventional radiographs and with surgery (if available).

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of wrist instability or wrist pain
* Previous medical examination
* Informed consent
* Must have a social security number

Exclusion Criteria:

* MR or CT contra-indications
* No prior surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
scapholunate diastasis (mm) | 1 day
  The distance between the scaphoid bone and the lunate bone will be measured during all maneuvers performed
Scapholunate angle | 1 day
  the variation in the scapholunate angle during the maneuvers performed will be assessed
Lunocapitate angle | 1 day
  the variation in the lunocapitate angle during the maneuvers performed will be assessed
Posterior radio scaphoid angle | 1 Day
  The angle formed between the posterior most point of the scaphoid in the sagittal plane and the ventral and dorsal rims of the distal radius will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Alain Blum, MD, PhD, Study Director — Central Hospital, Nancy, France
Locations (1):
- CentralHNF, Nancy, Lorraine, France

REFERENCES:
- [Background] Gondim Teixeira PA, Gervaise A, Louis M, Lecocq S, Raymond A, Aptel S, Blum A. Musculoskeletal wide detector CT: principles, techniques and applications in clinical practice and research. Eur J Radiol. 2015 May;84(5):892-900. doi: 10.1016/j.ejrad.2014.12.033. Epub 2015 Jan 17. PMID 25656096
- [Background] Garcia-Elias M, Alomar Serrallach X, Monill Serra J. Dart-throwing motion in patients with scapholunate instability: a dynamic four-dimensional computed tomography study. J Hand Surg Eur Vol. 2014 May;39(4):346-52. doi: 10.1177/1753193413484630. Epub 2013 Apr 8. PMID 23571486
- [Background] Halpenny D, Courtney K, Torreggiani WC. Dynamic four-dimensional 320 section CT and carpal bone injury - a description of a novel technique to diagnose scapholunate instability. Clin Radiol. 2012 Feb;67(2):185-7. doi: 10.1016/j.crad.2011.10.002. Epub 2011 Dec 3. No abstract available. PMID 22137722
- [Background] Troupis JM, Amis B. Four-dimensional computed tomography and trigger lunate syndrome. J Comput Assist Tomogr. 2013 Jul-Aug;37(4):639-43. doi: 10.1097/RCT.0b013e31828b68ec. PMID 23863544
- [Derived] Orkut S, Gillet R, Granero J, Hossu G, Douis N, Athlani L, Blum A, Gondim Teixeira PA. Assessment of Scapholunate Instability on 4D CT Scans in Patients with Inconclusive Conventional Images. Radiology. 2023 Sep;308(3):e230193. doi: 10.1148/radiol.230193. PMID 37698480